CLINICAL TRIAL: NCT02741973
Title: Yoga in School Sports - a Non-randomized Controlled Pilot Study in Germany
Brief Title: Yoga in School Sports - a Pilot Study in Germany
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Andreas Michalsen, Prof. Dr., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SchoolYoga
Record Dates: First submitted 2016-03-23; First posted 2016-04-18 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Yoga; Stress
Keywords: Yoga; Stress; Adolescents; School; Children
MeSH Terms: interventions — Yoga

ARMS (2):
- Yoga (Experimental): Students have 10 weeks yoga instead of school sport.
  Interventions: Other: Yoga
- School sport (Active Comparator): Students have 10 weeks regular school sport.
  Interventions: Other: School sport

INTERVENTIONS:
Other: Yoga
  Arms: Yoga
Other: School sport
  Arms: School sport

SUMMARY:
The aim of this trial is a first evaluation of the effectiveness of yoga as alternative for school sports to evaluate potential effects in stress reduction and concomitant psychological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Students of Berlin Oberstufenzentrum (OSZ) aged 17-27 years
* Written consent (with parents at underage (17 years)

Exclusion Criteria:

* Severe chronic or acute diseases
* Pregnancy or lactation
* Immobility or restriction for gymnastic exercises because of orthopedic, neurological or other medical reasons
* Participation in another study

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cohen Perceived Stress Scale (CPS) | Change in CPS from Baseline to 10 weeks

SECONDARY OUTCOMES:
Cohen Perceived Stress Scale (CPS) | Change in CPS from Baseline to 6 months
WHO-5 questionaire (quality of life) | Baseline, 10 weeks, 6 months
Hospital Anxiety and Depression (HADS) | Baseline, 10 weeks, 6 months
Profile of Mood States (POMS) | Baseline, 10 weeks, 6 months
Visual analogue scales (VAS) for general pain, headache, shoulder and neck tension, fatigue, sleep quality | Baseline, 10 weeks, 6 months
D2 Test of Attention | Baseline, 10 weeks, 6 months
  The d2 Test of Attention is a neuropsychological paper-and-pencil test of selective and sustained attention. Participants have to cross out any letter "d" with two marks around above it or below it in any order. Surrounding distractors are similar to the target stimulus, e.g. a "p" with two marks.
Yoga Self-Efficacy Scale | Baseline, 10 weeks, 6 months
Overall assessment of efficacy and tolerability (Likert scales) | Baseline, 10 weeks, 6 months

OTHER OUTCOMES:
Heart rate variability | Baseline, 10 weeks, 6 months
Qualitative interviews in focus groups | 5 weeks, 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany